CLINICAL TRIAL: NCT02149979
Title: Closure of Skin Incision Using CO2 Laser
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avraham Katzir (Other)
Responsible Party: Sponsor-Investigator, Avraham Katzir, Head of the applied physics group, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Katzir #1
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Wound
Keywords: Incision; Wound Closure; Laser Tissue Soldering
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temperature Controlled Laser Soldering (Experimental): Efficacy and safety of Temperature Controlled Laser Soldered wound incisions closure
  Interventions: Device: Temperature Controlled Laser Soldering

INTERVENTIONS:
Device: Temperature Controlled Laser Soldering — This study had a prospective within-subject design. Patients allocated to laparoscopic cholecystectomy procedure were enrolled. After the completion of the laparoscopic cholecystectomy surgical procedure, 4 trocar port sites were randomly either sutured or laser soldered by employing the temperature-controlled laser soldering system.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using Temperature Controlled Laser Soldering System for soft tissue bonding.

DETAILED DESCRIPTION:
Skin incisions can be closed by a variety of method which create temporary approximation of the wound edges until natural healing process ensue and reach a phase, where it is closed and can sustain the daily tensile forces.

The wound closure devices include sutures, staples, tapes, tissue adhesives. The Applied Physics group at the Tel Aviv University has developed a Temperature Controlled CO2 Laser Soldering system for soft tissue bonding.

This system includes features that make laser soldering suitable for clinical use. The Temperature Controlled Laser Soldering System is composed of CO2 fiberoptic laser device, Infrared fiber-optic radiometer, a computerized temperature control program, propriety grip device (Clamps) and concentrated Human Albumin as a soldering agent.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age 18-65.
* Subject is scheduled for laparoscopic cholecystectomy surgery.
* Subject able to comprehend and sign informed consent for participation in this study.
* Ability to comply with the study procedures and follow-up visits

Exclusion Criteria:

* Subject has a history of hypertrophic or keloid scar formation
* Subject is a pregnant and/or nursing woman
* Subject has a known allergy to blood products
* Subject is suffering from a bleeding disorders or using anticoagulant medications
* Subject is suffering from hepatic or renal disorder
* Subject is suffering from rheumatic and / or collagen disorder
* Subject is using steroids
* Subject is suffering from immunosuppressive disorder
* Subject is suffering from Ischemic Heart Disease (IHD)
* Subject is suffering from neoplastic disorder
* Subject who has had an active illness within 4 weeks of study enrollment
* Subject is participating in another study for an investigational drug and/or device within 3 months of study enrollment
* Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Primary study endpoint will be to establish the safety of using the Temperature Controlled Laser Soldering System for skin bonding and wounds closure. Safety will be established by paucity of serious adverse events and adverse events. | 3 months

SECONDARY OUTCOMES:
Re-intervention: A subject is scored a success (1) if he had No Re-intervention by 3 months; otherwise he is scored a failure (0). | 3 months
Wound dehiscence of at least 50% of wound length | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Doron Kopelman, MD, Principal Investigator — Department of Surgery B, "HaEmek" Medical Center, Afula,; Abraham Katzir, PhD, Study Chair — The applied physics group, Tel Aviv University; David Simhon, MD, PhD, Study Director — The applied physics group, Tel Aviv University
Locations (2):
- Israel (2):
  - Department of Surgery B, "HaEmek" Medical Center, Afula
  - Haemek Medical Center, Afula

REFERENCES:
- [Background] Simhon D, Halpern M, Brosh T, Vasilyev T, Ravid A, Tennenbaum T, Nevo Z, Katzir A. Immediate tight sealing of skin incisions using an innovative temperature-controlled laser soldering device: in vivo study in porcine skin. Ann Surg. 2007 Feb;245(2):206-13. doi: 10.1097/01.sla.0000232554.13719.10. PMID 17245173
- [Background] Simhon D, Brosh T, Halpern M, Ravid A, Vasilyev T, Kariv N, Katzir A, Nevo Z. Closure of skin incisions in rabbits by laser soldering: I: Wound healing pattern. Lasers Surg Med. 2004;35(1):1-11. doi: 10.1002/lsm.20074. PMID 15278922
- [Background] Brosh T, Simhon D, Halpern M, Ravid A, Vasilyev T, Kariv N, Nevo Z, Katzir A. Closure of skin incisions in rabbits by laser soldering II: Tensile strength. Lasers Surg Med. 2004;35(1):12-7. doi: 10.1002/lsm.20073. PMID 15278923
- [Background] Simhon D, Ravid A, Halpern M, Cilesiz I, Brosh T, Kariv N, Leviav A, Katzir A. Laser soldering of rat skin, using fiberoptic temperature controlled system. Lasers Surg Med. 2001;29(3):265-73. doi: 10.1002/lsm.1118. PMID 11573230